CLINICAL TRIAL: NCT02390830
Title: Falls Prevention and Balance Rehabilitation in Multiple Sclerosis: a Bi-centre Randomized Control Trial
Brief Title: Falls Prevention and Balance Rehabilitation in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT_SM_Falls
Record Dates: First submitted 2015-03-06; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention (Experimental): Participants in the intervention group received at least 25-45' of balance treatment. The balance treatments were aimed at improving participants' control of the position and movement of the center of mass and body segments during static, dynamic and transitional tasks.
  Interventions: Other: Falls Prevention
- Control (Active Comparator): Participants in the control group were treated to reduce limitations at body function and activity levels, while treatment for balance disorders was restricted to a maximum of 10' per session. Treatment mainly focused on increasing range of joints motion, reducing of muscle contractures and strength training.
  Interventions: Other: Reduction of limitations at body function and activity levels

INTERVENTIONS:
Other: Falls Prevention
  Arms: Intervention
Other: Reduction of limitations at body function and activity levels
  Arms: Control

SUMMARY:
Background. Balance disorders and falls are common in People with Multiple Sclerosis (PwMS) Objective: Our hypothesis was that PwMS treated for balance disorders would reduce balance disorders and frequency of falls.

Methods: A bi-centre randomised Rater-blinded controlled trial. Participants in both groups received 20 treatment sessions. Participants in the intervention group received treatment aimed at improving control of the position and movement of the centre of mass and body segments. Participants in the control group received treatments to reduce limitations at activity and body function level.

Group allocation was done by an independent clinician by a randomization list made before the beginning of the study. Group allocation was kept concealed throughout the study and participants were not aware of group assignment.

Data was analyzed according to a preplanned protocol by using an intention to treat approach.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Multiple Sclerosis Must be able to walk (also with aid) for 6m Must be able to maintain standing position with open eyes for at least 30".

Exclusion Criteria:

Must not be able to maintain monopodalic-standing position for 10", Must not be able to to maintain tandem position for 30", cognitive disorders hampering the execution of the exercises/assessment.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Frequency of fallers at 2 and 4 months | baseline, then participants were followed for the duration the outpatient treatment protocol, an average of 8 weeks, and at follow up 2 months after the end of the treatment protocol